CLINICAL TRIAL: NCT00014482
Title: Music Therapy for Distress During Autologous Stem Cell Transplantation: A Randomized Trial
Brief Title: Music Therapy to Ease Pain and Emotional Distress in Patients With Hematologic Cancer Who Are Undergoing High-Dose Therapy and Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized
Other Study IDs: 00-134; CDR0000068547 (Registry Identifier: PDQ (Physician Data Query)); NCI-G01-1934
Record Dates: First submitted 2001-04-10; First posted 2003-01-27 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Anxiety Disorder; Chronic Myeloproliferative Disorders; Depression; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Pain
Keywords: anxiety disorder; depression; pain; recurrent adult Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; primary myelofibrosis; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Anxiety Disorders; Myeloproliferative Disorders; Depression; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Pain; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Primary Myelofibrosis; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Analgesia; Psychiatric Rehabilitation

INTERVENTIONS:
Procedure: pain therapy
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Music therapy may be effective in relieving pain and emotional distress in patients who are undergoing cancer therapy.

PURPOSE: Randomized trial to determine the effectiveness of music therapy to ease pain and emotional distress in patients with hematologic cancer who are undergoing high-dose therapy and stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effects of music therapy vs no music therapy on depression and anxiety in patients with hematologic malignancies undergoing high-dose therapy and autologous stem cell transplantation.
* Compare the effects of these regimens on mood, mucositis pain, pain interference, need for analgesic medication, and length of hospital stay of these patients.
* Compare the immediate effects of these regimens on mood in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to whole body or whole lymphatic irradiation (yes vs no) and diagnosis (non-Hodgkin's lymphoma vs Hodgkin's lymphoma vs myeloma/amyloidosis). Patients are randomized to one of two arms.

* Arm I: Patients receive individualized music therapy over 20-30 minutes beginning on day 0 and continuing over 16 days for a maximum of 12 sessions during high-dose therapy and autologous stem cell transplantation.

Patients complete a Profile of Mood States (POMS) quality of life and pain questionnaire on days -2, 0, 1, 4, 7, 10, 13, and 16.

* Arm II: Patients receive standard psychosocial support during high-dose therapy and autologous stem cell transplantation. Patients complete POMS and mucositis pain questionnaires as in arm I.

PROJECTED ACCRUAL: A total of 80 patients (40 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a hematologic malignancy

  * No leukemia
* Planned high-dose therapy and autologous stem cell transplantation (HDT/ASCT) at Memorial Sloan-Kettering Cancer Center

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No prior HDT/ASCT

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-12; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barrie R. Cassileth, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States